CLINICAL TRIAL: NCT04030312
Title: Effectiveness of Donor Human Milk Supplementation Compared to Infant Formula for the Treatment of Hypoglycemia in the Breastfed Infant in the Normal Newborn Nursery
Brief Title: Effectiveness of Donor Human Milk Supplementation for the Treatment of Hypoglycemia in the Breastfed Infant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0119-19-EP
Record Dates: First submitted 2019-04-11; First posted 2019-07-23 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Neonatal Hypoglycemia
Keywords: neonatal; newborn; hypoglycemia; human milk; breastfed; donor milk
MeSH Terms: conditions — Hypoglycemia; Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Infant Formula (Active Comparator): Infants in this randomized treatment arm will receive bottle supplementation of up to 15 milliliters of standard 20 calorie-per-ounce infant formula up to two times during the duration of the study to treat hypoglycemia.
  Interventions: Dietary Supplement: Bottle Supplementation--Standard Infant Formula
- Commercially-Sterilized Donor Human Milk (Experimental): Infants in this randomized treatment arm will receive bottle supplementation of up to 15 milliliters of 20 calorie-per-ounce commercially-sterilized donor human milk up to two times during the duration of the study to treat hypoglycemia.
  Interventions: Dietary Supplement: Bottle Supplementation--Commercially-Sterilized Donor Human Milk

INTERVENTIONS:
Dietary Supplement: Bottle Supplementation--Commercially-Sterilized Donor Human Milk — Supplementation by bottle with 20-calorie-per-ounce commercially-sterilized donor human milk (up to 15 ml, up to two times) for infants meeting hypoglycemia criteria and randomized to this treatment arm.
  Arms: Commercially-Sterilized Donor Human Milk
Dietary Supplement: Bottle Supplementation--Standard Infant Formula — Supplementation by bottle with 20-calorie-per-ounce standard infant formula (up to 15 ml, up to two times) for infants meeting hypoglycemia criteria and randomized to this treatment arm.
  Arms: Standard Infant Formula

SUMMARY:
The purpose of this study is to compare if newborn infant hypoglycemia can be improved with bottle supplementation of commercially-sterilized donor human milk compared to standard infant formula. Hypothesis is that supplementation with commercially-sterilized donor human milk will improve hypoglycemia and limit formula use in exclusively breastfed infants.

DETAILED DESCRIPTION:
Enrolled infant participants will receive a maximum of two bottle feeding supplementations (of their designated treatment arm for either 20 calorie-per-ounce commercially-sterilized donor human milk OR 20-calorie-per-ounce standard infant formula) as treatment if they meet hypoglycemia criteria. Infant participants will complete the study if 1) they have received two bottle feeding supplementations for treatment of hypoglycemia, 2) they only received one bottle supplementation and hypoglycemia resolved, 3) if the medical teams deems the infants requires a higher level of care for their hypoglycemia (example: admission to the newborn intensive care unit for intravenous fluids with dextrose).

ELIGIBILITY:
Mother-infant pairs will be consented for participation via informed written consent.

Inclusion Criteria:

* Mother/infant dyads deliverying at Nebraska Medicine hospital (Omaha, NE, USA).
* Infant in the normal newborn nursery, born greater than or equal to 36 weeks gestational age.
* Infant with blood glucose after delivery of < 40 milligrams/deciliter within the first four hours of life OR blood glucose levels less than 45 milligrams/deciliter after four hours of life
* Deliverying mother plans to exclusively breastfeed.

Exclusion Criteria:

* Infants born and directly admitted to the newborn intensive care unit
* Infants with known congenital abnormality or known inborn error of metabolism that influences growth and metabolic outcomes
* Infants deemed ward of state
* Mothers who do not plan to exclusively breastfeed at time of delivery
* Mothers less than 19 years of age

Ages: 1 Minute to 72 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2023-04-10 (Actual)

PRIMARY OUTCOMES:
Effectiveness of Resolving Neonatal Hypoglycemia: Blood glucose levels | Blood glucose levels will be monitored within 60 minutes of initiating a feeding. Overall outcomes for each treatment arm will be compared at the completion of the study for all enrolled participants.
  To compare the effectiveness of commercially-sterilized donor human milk bottle supplementation for the treatment of hypoglycemia in the breastfed infant in the normal newborn nursery compared to bottle supplementation with standard infant formula.

SECONDARY OUTCOMES:
Exclusive Breastfeeding Duration | Families of consented participants will be contacted when the enrolled infant is 6 months old.
  To assess if donor human milk supplementation (when compared to formula supplementation) impacts rate of exclusive breastfeeding during the first 6 months of life.
Parenteral Satisfaction of Infant Feeding: Parenteral satisfaction surveys | Parenteral satisfaction surveys will be completed prior to mother's hospital discharge (within 72 hours following delivery).
  To compare if donor human milk supplementation (when compared to formula supplementation) improves parental satisfaction related to infant feeding during post-partum hospitalization.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa K Thoene, RD, PhD, Principal Investigator — Nebraska Medicine
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No